CLINICAL TRIAL: NCT01919788
Title: Intracellular Counter-regulatory Mechanisms Following Low Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Thomas Schmidt Voss, MD, University of Aarhus
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: VEK journal nr.: M-2013-113-13; VEK Journal nr. M-2013-113-13 (Other: VEK)
Record Dates: First submitted 2013-08-05; First posted 2013-08-09 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus Type I; Hypoglycemia
Keywords: Diabetes Mellitus Type I; Hypoglycemia; Counter-regulatory mechanisms
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Insulin; Glucose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): No insulin administered. Instead of insulin infusion, a small amount of saline is administered to keep the subject blinded.
  Three muscle biopsies and two fat biopsies will be obtained. A palmitic acid tracer will be given to estimate fatty acid metabolism. Forearm pletysmography will be performed twice.
  Interventions: Other: Saline
- Insulin (Experimental): Insulin (Insuman Rapid) is administered once as a bolus of 0,1 IU/kg. Three muscle biopsies and two fat biopsies will be obtained. A palmitic acid tracer will be given to estimate fatty acid metabolism Forearm pletysmography will be performed twice
  Interventions: Drug: Insulin (Insuman Rapid)
- Insulin and glucose (Experimental): Insulin (Insuman rapid) is administered once as a bolus injection of 0,1 IU/kg and glucose is given at the same time to avoid hypoglycemia in this arm.
  Three muscle biopsies and to fat biopsies is obtained. A palmitic acid tracer is given to estimate fatty acid metabolism Forearm pletysmography will be performed twice
  Interventions: Drug: Insulin (Insuman Rapid); Drug: Glucose

INTERVENTIONS:
Drug: Insulin (Insuman Rapid)
  Arms: Insulin; Insulin and glucose
Drug: Glucose
  Arms: Insulin and glucose
Other: Saline
  Arms: Control

SUMMARY:
Diabetes mellitus type I (DMI) is characterized by lack of endogenous insulin and these patients are 100% dependent on insulin substitution to survive. Diabetes mellitus type II (DMII) is characterized by reduced insulin sensitivity and sometimes also reduced insulin production, thus patients with DMII might also be dependent on insulin substitution.

Insulin is produced in- and secreted from the pancreas when blood glucose concentration rises during- and after a meal. Insulin increases cellular uptake of glucose leading to lower blood glucose concentration. Substitution with insulin is/can be necessary in DM, but at the same time it induces the risk of hypoglycemia. This makes treatment with insulin a balancing act between hyper- and hypoglycemia.

A hypoglycemic episode is a dreaded consequence of insulin overdosing, and also a very frequent reason for hospital admission in patients with DM. Examples of hypoglycemic symptoms may be; shaking, a sense of hunger, sweating, irritability progressing to lack of relevant cerebral responses and eventually coma, convulsions and possibly death. People with diabetes lose the ability to sense of low blood glucose with time, because of a lack of appropriate counter-regulatory responses, hereby increasing the risk of severe hypoglycemia. Understanding normal physiologic counter regulatory mechanisms during hypoglycemia is of major importance to patients with DM and has the potential to change medical treatment in diabetes, to reduce the risk of hypoglycemia.

Hypothesis: Hypoglycemia counteracts insulin signaling via hormone-dependent intracellular counter-regulatory mechanisms, involving phosphorylation of specific signaling proteins.

Aim: To define counter-regulatory mechanisms in muscle- and fat tissue during hypoglycemia, and to investigate the effect of insulin on lipid metabolism in healthy- and type I diabetic subjects.

ELIGIBILITY:
* BMI > 19 and < 26
* Written Consent

Exclusion Criteria:

* Epilepsy
* Cardiac arrythmia
* Ischemic heart disease
* Other medical illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Insulin and growth hormone signalling, expressed as CHANGE in phosphorylation of intracellular target proteins and mRNA expression of target genes in muscle- and fat-tissue. | Biopsies obtained on each study day (arm). Muscle biopsies: time (t)= -30min, t= 30min and t= 75min. Fat biopsies: t= 30min and t= 75min
  Change in phosphorylation of target proteins and mRNA expression of target genes assessed with western blotting technique.

SECONDARY OUTCOMES:
Intracellular markers of lipid metabolism in muscle- and fat tissue biopsies. | Biopsies obtained on each study day (arm). Muscle biopsies: time (t)= -30min, t= 30min and t= 75min. Fat biopsies: t= 30min and t= 75min
  Assessed by Western blotting.
Metabolism. | measured twice on each study day (arm) at t= -30-0 min. and t= 50-80 min.
  Assessment of glucose metabolism by forearm pletysmography and heated hand technique (duration of pletysmography = 30 min.)
Ghrelin | Measured at t = -30min., t=0min, t=15min, t= 30min., t=45min., t=60min., t= 75min., t=90min. and t=105min. on each study day (arm)
Metabolism | once per study day (arm): t 45min - 105min.
  A palmitic acid tracer will be given once per trial day to estimate fatty acid metabolism. Duration 1 hour.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, MD, Study Chair — Aarhus University / Aarhus University Hospital; Thomas Voss, MD, Principal Investigator — Aarhus University / Aarhus University Hospital
Locations (1):
- Institute of Clinical Medicine, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Derived] Voss TS, Vendelbo MH, Kampmann U, Hingst JR, Wojtaszewski JFP, Svart MV, Moller N, Jessen N. Acute Hypoglycemia in Healthy Humans Impairs Insulin-Stimulated Glucose Uptake and Glycogen Synthase in Skeletal Muscle: A Randomized Clinical Study. Diabetes. 2017 Sep;66(9):2483-2494. doi: 10.2337/db16-1559. Epub 2017 Jun 8. PMID 28596236
- [Derived] Voss TS, Vendelbo MH, Kampmann U, Pedersen SB, Nielsen TS, Johannsen M, Svart MV, Jessen N, Moller N. Effects of insulin-induced hypoglycaemia on lipolysis rate, lipid oxidation and adipose tissue signalling in human volunteers: a randomised clinical study. Diabetologia. 2017 Jan;60(1):143-152. doi: 10.1007/s00125-016-4126-x. Epub 2016 Oct 12. PMID 27734104